CLINICAL TRIAL: NCT04382924
Title: A Randomized Open Label Phase 2b/3 Study of the Safety and Efficacy of NP-120 (Ifenprodil) for the Treatment of Hospitalized Patient With Confirmed COVID-19 Disease
Brief Title: Safety and Efficacy of NP-120 (Ifenprodil) for the Treatment of Hospitalized Patient With Confirmed COVID-19 Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Algernon Pharmaceuticals (Industry)
Collaborators: Novotech (Australia) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGN120-3
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: COVID
MeSH Terms: interventions — ifenprodil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm A (Experimental): NP-120 (Ifenprodil) 20 mg TID + Standard of Care
  Interventions: Drug: NP-120 (Ifenprodil)
- Control Arm (No Intervention): Standard of Care only
- Treatment Arm B (Experimental): NP-120 (Ifenprodil) 40 mg TID + Standard of Care
  Interventions: Drug: NP-120 (Ifenprodil)

INTERVENTIONS:
Drug: NP-120 (Ifenprodil) — Ifenprodil, 20 mg TID Ifenprodil, 40 mg TID
  Arms: Treatment Arm A; Treatment Arm B

SUMMARY:
The purpose of this adaptive trial is to determine the clinical efficacy of Ifenprodil in the treatment of patients infected with COVID-19. This Protocol is largely based on the recommendations of the World Health Organization (WHO) R&D Blueprint Clinical Trials Expert Group COVID-19 Therapeutic Trial Synopsis, and associated Master Protocol.

The choice of the primary outcome measure will be determined by a pilot study of the first 150 subjects. Subject clinical status (on a 7-point ordinal scale) at day 15 in treatment versus the control group is the default primary endpoint.

DETAILED DESCRIPTION:
NP-120 (Ifenprodil) is an N-methyl-D-Aspartate (NDMA) inhibitor that is specific for the NR2B subunit of the NMDA Receptor. The NMDA receptor, and specifically the NR2B subunit, is involved in glutamate signaling, and is expressed on both neutrophils and T cells. In the case of neutrophils, activation of the NMDA receptor can (1) result in expression of CD11b which targets neutrophils via ICAM-1 to areas of inflammation, and (2) trigger the autocrine release of glutamate. In the case of T-cells, activation of T cells via glutamate can cause (1) T cell proliferation and, (2) the release of cytokines. The activation of T cells and cytokine release can be blocked in vitro by the addition of Ifenprodil. As such it could be a potent anti-inflammatory agent.

Ifenprodil was discovered by a genome wide RNAi assay to uncover gene targets associated with cytoprotective activity against highly pathogenic H5N1 influenza, specifically by preserving cell viability in vitro. When tested in a murine model of H5N1, the drug at clinically relevant doses: (1) improved survivability from 0% at day 6 to 40% day 14 post-infection, (2) the drug significantly reduced edema and lung injury score and (3) reduced infiltrating T cells, neutrophils and NK cells and attenuated the 'cytokine storm'. The mortality rate of H5N1 in humans is >50%, whereas the mortality rate of COVID-19 infected patients is < 5%, and both viruses cause acute lung injury and share similar pulmonary pathologies. NP-120 has also been shown to mediate anti-inflammatory responses and reduce pulmonary fibrosis in a murine model of idiopathic pulmonary fibrosis, a complication which can occur after a respiratory virus infection.

Based on the fact that H5N1 has a significantly higher mortality rate than COVID-19 but still shares similar lung pathologies, Algernon Pharmaceuticals believes Ifenprodil could reduce lung injury associated with COVID-19 infection, thereby improving lung function and accelerating patient recovery.

The purpose of this Phase 2b/3 trial is to determine the safety and efficacy of NP-120 in the treatment of COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged ≥18 years of age
2. Confirmed coronavirus infection

   1. Positive real-time fluorescence polymerase chain reaction of the patient's respiratory or blood specimens for COVID-19 nucleic acid
   2. Viral gene sequences in respiratory or blood specimens that are highly homologous to COVID-19
   3. Any other diagnostic test accepted by local regulatory authorities
3. Must be hospitalized and requiring supplemental oxygen, or on non-invasive ventilation or high flow oxygen devices (Score of 4 or 5 on WHO Ordinal Clinical Scale)
4. Female subjects of childbearing potential who are sexually active with a non-sterilized male partner must use at least 1 highly effective method of contraception (e.g. oral contraceptives, intrauterine device, diaphragm plus spermicide) from the time of screening and must agree to continue using such precautions for 90 days after the final dose of study drug(s)
5. Non-sterilized males who are sexually active with a female partner of childbearing potential must use condom plus spermicide from day 1 through 90 days after receipt of the last dose of study drug(s)
6. Subjects (or reasonable legal designate) must have the capacity to understand, sign and date a written, informed consent form and any required authorization prior to initiation of any study procedures

Exclusion Criteria:

1. Patients with vasodilatory shock, orthostatic hypotension, hypotension, or tachycardia at screening/baseline
2. Patients experiencing cerebral hemorrhage or cerebral infarction at baseline
3. ALT/AST > 5 times the upper limit of normal; Child-Pugh Score 10 to 15
4. Stage 4 severe chronic kidney disease or requiring dialysis (i.e. eGFR < 30)
5. Patients on mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
6. Patients taking droxidopa
7. Pregnant and lactating women and those planning to get pregnant
8. Known or suspected allergy to the trial drug or the relevant drugs given in the trial
9. Presence of other disease that may interfere with testing procedures or in the judgement of the Investigator may interfere with trial participation or may put the patient at risk when participating in this trial
10. Know inability of patient to comply with the protocol for the duration of the study
11. Involvement in a clinical research study within 4 weeks prior to screening and/or prior enrollment in the study or plan to participate in another interventional clinical trial during the study period. Participation in observational registry studies is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - Westchester Research Center, Miami, Florida
  - Affinity Health - Loretto Hospital, Chicago, Illinois
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Promedica Health: Toledo Hospital and BayPark Hospital, Toledo, Ohio
- Australia (2):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Melbourne Hospital, Parkville, Victoria
- Philippines (3):
  - Makati Medical Center, Manila
  - Philippine General Hospital, Manila
  - Lung Center of the Philippines, Quezon City
- National Institute of Infectious Diseases, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
Started | 52 | 56 | 60
Completed | 44 | 46 | 48
Not Completed | 8 | 10 | 12
Not completed — Death | 2 | 5 | 4
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Transferred to other hospital/declined in person visits | 0 | 1 | 1
Not completed — Withdrawal by Subject | 6 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm | Total
Number analyzed (Participants) | 52 | 56 | 60 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 36 | 36 | 110
  >=65 years | 14 | 20 | 24 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (13.1) | 58.5 (14.5) | 59.7 (12.9) | 58.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 27 | 21 | 68
  Male | 32 | 29 | 39 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 7 | 13
  Not Hispanic or Latino | 49 | 52 | 53 | 154
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 16 | 18 | 18 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 35 | 35 | 41 | 111
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Romania | 29 | 29 | 30 | 88
  United States | 7 | 10 | 12 | 29
  Philippines | 15 | 17 | 18 | 50
  Australia | 1 | 0 | 0 | 1
Patient clinical status on WHO 7 point ordinal scale [Mean (Standard Deviation); unit: scores on a scale] | 4.23 (0.425) | 4.25 (0.548) | 4.25 (0.437) | 4.24 (0.471)

OUTCOME MEASURES:

1. Primary Outcome: Patient Clinical Status (on the WHO 7-point Ordinal Scale) at Day 15 in IP Versus SOC Control Group Patients:
Description: 1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or ECMO
  7. Death
Time Frame: Day 15
Population: Analysis performed on the number of patients with WHO-7 data
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
Number analyzed (Participants) | 46 | 44 | 48
Participants
  1. Not hospitalized no limitations on activities | 10 | 9 | 18
  2. Not hospitalized but limitations on activities | 7 | 9 | 2
  3. Hospitalized not requiring supplemental O2 | 13 | 13 | 16
  4. Hospitalized and requires supplemental O2 | 13 | 8 | 7
  5. Hospitalized and on non-invasive ventilation or high flow O2 | 1 | 1 | 1
  6. Hospitalized and on mechanical ventilation or ECMO | 2 | 1 | 2
  7. Death | 0 | 3 | 2
Statistical Analysis 1: Comparison: Treatment Arm A vs Treatment Arm B vs Control Arm; Test type: Superiority; p < 0.025, Chi-squared; Odds Ratio, log = 0.0001

2. Secondary Outcome: Status on an Ordinal Scale Assessed Daily While Hospitalized and on Days 15 and 28 in IP Versus Control Group Patients
Description: WHO status of subjects at timepoints from baseline to day 28
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or ECMO
  7. Death
Time Frame: Days 1 through 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
Number analyzed (Participants) | 52 | 56 | 60
scores on a scale
  Baseline | 4.23 (0.425) | 4.25 (0.548) | 4.25 (0.427)
  Day 3 | 4.22 (0.503) | 4.22 (0.718) | 4.29 (0.7063)
  Day 5 | 4.12 (0.627) | 4.14 (0.917) | 4.18 (0.819)
  Day 8 | 3.89 (0.767) | 4.02 (1.012) | 4.04 (0.988)
  Day 11 | 3.87 (0.777) | 4.09 (1.156) | 3.97 (1.098)
  Day 15 | 2.87 (1.343) | 2.95 (1.628) | 2.96 (1.665)
  Day 28 | 1.59 (1.384) | 1.80 (1.608) | 1.73 (1.730)

3. Secondary Outcome: NEWS Assessed Days 3, 5, 8 ,11 Daily While Hospitalized and on Days 15 and 29 in IP Versus Control Group Patients
Description: National Early Warning Score assessed between baseline and Day 29 on subjects in 20, 40 mg TID NP-120 arms versus control group
  The National Early Warning Score (NEWS) scale is a composite of 7 physiological parameters: Respiration Rate (per minute),Oxygen Saturations (%), Any Supplemental Oxygen, Temperature (°C), Systolic BP (mmHg), Heart Rate (per minute), Level of Consciousness. The aggregate results from all 7 physiological parameters are used to obtain the NEW Score., ranging from 0 - 20. Higher values reflect a worse outcome.
Time Frame: Days 3, 5, 8, 11, 25, 29
Population: NEWS score collected on patients currently hospitalized, or returning for follow up visits
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
Number analyzed (Participants) | 52 | 56 | 60
scores on a scale
  Baseline | 4.7 (1.83) | 4.5 (1.58) | 4.5 (1.51)
  Day 3: number analyzed (Participants) | 51 | 53 | 55
  Day 3 | 4.2 (1.90) | 3.7 (1.60) | 4.4 (1.91)
  Day 5: number analyzed (Participants) | 50 | 49 | 54
  Day 5 | 3.8 (2.04) | 3.3 (1.95) | 3.7 (1.99)
  Day 8: number analyzed (Participants) | 46 | 40 | 45
  Day 8 | 3.5 (2.33) | 3.1 (2.04) | 3.0 (2.51)
  Day 11: number analyzed (Participants) | 38 | 30 | 34
  Day 11 | 3.0 (2.21) | 3.0 (2.60) | 3.2 (2.39)
  Day 15: number analyzed (Participants) | 46 | 39 | 44
  Day 15 | 2.4 (2.85) | 1.8 (2.38) | 1.8 (2.37)
  Day 29: number analyzed (Participants) | 36 | 39 | 40
  Day 29 | 1.1 (1.97) | 1.4 (2.10) | 1.3 (2.11)

4. Secondary Outcome: Rate of Mechanical Ventilation in IP Versus Control Group Patients
Description: Rate of mechanical ventilation in 20 and 40 mg TID NP-120 versus control group
Time Frame: Up to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
Number analyzed (Participants) | 52 | 56 | 60
Participants | 5 | 2 | 4

5. Secondary Outcome: Duration of Mechanical Ventilation (if Applicable) in IP Versus Control Group Patients
Description: Duration of mechanical ventilation in 20 and 40 mg TID subjects versus control who experience mechanical ventilation
Time Frame: Up to day 28
Measure: Number; unit: participants
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
Number analyzed (Participants) | 5 | 2 | 4
participants
  < 6 hours | 0 | 1 | 0
  >= 12 hours but < 24 hours | 0 | 0 | 0
  >= 24 hours but <72 hours | 1 | 0 | 0
  >=72 hours but <120 hours | 0 | 1 | 1
  >= 120 hours | 3 | 0 | 2
  Ongoing at time of EOS (>= 24 hours but <72 hours | 1 | 0 | 1

6. Secondary Outcome: Duration of Supplemental Oxygen in IP Versus Control Group Patients
Description: Duration in patients only receiving supplemental oxygen in IP versus control group up to Day 29
Time Frame: Up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
Number analyzed (Participants) | 46 | 48 | 52
Participants
  < 6 hours | 0 | 0 | 0
  >= 12 hours but < 24 hours | 0 | 1 | 0
  >= 24 hours but < 72 hours | 4 | 4 | 5
  >= 72 hours but < 120 hours | 7 | 5 | 8
  >= 120 hours | 35 | 38 | 39

7. Secondary Outcome: Time to Return to Room Pressure (SpO2 > 94%) on Room Air
Description: Time to return to room pressure (SpO2 > 94%) on room air in patients in 20, 40 mg TID NP-120 groups versus control group with 94% blood oxygen levels at enrolment
  Time-to-event endpoints with competing risk were analysed for each dosing group using the Cumulative Incidence Function-CIF (KM) graphical display. Data represents the time (in Days) it took for all participants in the group to return to room pressure air (e.g. the time when the CIF curve hit 100%).
Time Frame: Up to Day 29
Measure: Number; unit: Days
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
Number analyzed (Participants) | 11 | 11 | 13
Days | 4 | 5 | 9

8. Secondary Outcome: Duration in ICU (if Applicable) in IP Versus Control Group Patients
Description: Duration of subject in ICU in 20 and 40 TID mg groups versus control group patients
Time Frame: Up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
Number analyzed (Participants) | 8 | 6 | 9
Participants
  >= 1 day but < 3 days | 0 | 0 | 0
  >= 3 days but < 7 days | 1 | 0 | 1
  >=7 days but < 14 days | 3 | 3 | 3
  >=14 days but < 21 days | 1 | 1 | 2
  >= 21 days | 2 | 2 | 2
  Ongoing at end of study | 1 | 0 | 1

9. Secondary Outcome: Rate of Mortality in IP Versus Control Group Patients
Description: Rate of Overall Mortality in 20, 40 mg TID groups versus control group
Time Frame: Up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
Number analyzed (Participants) | 52 | 56 | 60
Participants | 2 | 5 | 4

10. Secondary Outcome: Duration of Hospitalization in IP Versus Control Group Patients
Time Frame: Day 15, 28
Reporting Status: Not Posted

11. Secondary Outcome: Time to Discharge in IP Versus Control Group Patients
Time Frame: Day 15, 28
Reporting Status: Not Posted

12. Secondary Outcome: Effect on the Rate of Change of Partial Pressure of Oxygen (PaO2) and PaO2/FiO2 Ratio Taken at Baseline and Measured Once Daily up to 2 Weeks of Treatment in IP Versus Control Group Patients
Time Frame: Up to day 15, day 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 60
Arm/Group | Treatment Arm A | Treatment Arm B | Control Arm
All-Cause Mortality (participants affected / at risk) | 2/52 | 5/56 | 4/60
Serious Adverse Events (participants affected / at risk) | 2/52 | 6/56 | 5/60
Other Adverse Events (participants affected / at risk) | 36/52 | 35/56 | 30/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A (N=52) | Treatment Arm B (N=56) | Control Arm (N=60)
Cardiac Arrest (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Cardiopulmonary Failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Coagulation test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A (N=52) | Treatment Arm B (N=56) | Control Arm (N=60)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 4 (4)
Oral candidiasis (Infections and infestations) | 6 (6) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 5 (5) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 3 (3)
Hepatocellular injury (Hepatobiliary disorders) | 4 (5) | 5 (5) | 8 (8)
Vessel puncture site bruise (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 3 (3)
Intertrigo (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT04382924/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT04382924/SAP_001.pdf